CLINICAL TRIAL: NCT04566692
Title: A Multi-center, Single-Sequence, Open-label Study to Evaluate IGSC 20% Biweekly Dosing in Treatment-Experienced Subjects and Loading/Maintenance Dosing in Treatment-Naïve Subjects With Primary Immunodeficiency
Brief Title: A Study to Evaluate IGSC 20% Biweekly Dosing in Treatment-Experienced Participants and Loading/Maintenance Dosing in Treatment-Naïve Participants With Primary Immunodeficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GC1906
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Primary Immunodeficiency
Keywords: Immunologic Deficiency Syndromes; Immune System Diseases; Immunoglobulins
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immunologic Deficiency Syndromes; Immune System Diseases | interventions — gamma-Globulins; Caprylates

STUDY DESIGN:
Intervention Model Description: Single sequence crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IGSC 20%: Treatment-experienced Cohort (Experimental): Participants first received 16 weekly doses of IGSC 20% using a subcutaneous (SC) infusion pump from Week 0 to Week 15. Participants entering study on intravenous immune globulin (IVIG), IGSC 20% was dosed at 1.37 times the equivalent weekly dose and participants entering on subcutaneous immunoglobulin (SCIG) received the same milligram/kilogram (mg/kg) equivalent weekly dose as given prior to study entry, without using a dose adjustment factor (DAF). Participants then received 9 biweekly doses of IGSC 20 % (i.e, IGSC 20% every 2 weeks) using an SC infusion pump, with the first IGSC 20% dose administered at Week 16 and the final dose given at Week 32.
  Interventions: Biological: IGSC 20%
- IGSC 20%: Treatment-naïve Cohort (Experimental): Treatment-naïve participants received a loading dose of 150 mg/kg/day of IGSC 20% for 5 consecutive days (Week 0, Days 1 to 5) followed by weekly maintenance infusions of 150 mg/kg IGSC 20% starting Week 1 (Day 8) through Week 32. IGSC 20% infusion was administered using an SC infusion pump.
  Interventions: Biological: IGSC 20%

INTERVENTIONS:
Biological: IGSC 20% — SC infusion pump.
  Other Names: Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified

SUMMARY:
The purpose of the study is to determine whether biweekly (every 2 weeks) administration of Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified (IGSC 20%) produces a steady-state area under the concentration versus time curve (AUC) of total Immunoglobulin G (IgG) that is non-inferior to that produced by weekly administration of IGSC 20% in treatment-experienced participants with primary immunodeficiency (PI).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria only for Treatment-Experienced Participants

* Participants 18 years to 75 years (inclusive) at screening
* Participants with documented and confirmed pre-existing diagnosis of Primary Immunodeficiency (PI) with features of hypogammaglobulinemia requiring Immunoglobulin G (IgG) replacement therapy including but not limited to the following humoral-based immunodeficiency syndromes (example, X-linked agammaglobulinemia, common variable immunodeficiency), and combined immunodeficiency syndromes without lymphocytopenia (example, hyper immunoglobulin M immunodeficiency syndrome).
* Participants have not had an Serious bacterial infection (SBI) or been hospitalized for infection of any etiology (example, viral, fungal, parasitic) within the last 3 months prior to screening or during screening.
* Participants currently receiving IgG replacement therapy for ≥3 months via Intravenous (IV) or SC infusion. Participants receiving IVIG prior to study must receive a dosage of at least 200 mg/kg per infusion.
* Participants whose screening IgG trough levels must be ≥500 milligram per deciliter (mg/dL).
* Participants have signed an informed consent form.

Inclusion Criteria only for Treatment-Naïve Participants

* Participants 6 years to 75 years (inclusive) at screening.
* Participants with documented and confirmed diagnosis of PI with features of hypogammaglobulinemia requiring IgG replacement therapy including but not limited to the following humoral-based immunodeficiency syndromes (example, X-linked agammaglobulinemia, common variable immunodeficiency), and combined immunodeficiency syndromes without lymphocytopenia (example, hyper immunoglobulin M immunodeficiency syndrome).
* Participants have never received IgG replacement treatment (ie, no prior immune globulin replacement therapy).
* Participants whose screening IgG level must be ≤400 mg/dL.
* Participants do not have an SBI nor requires hospitalization for infection of any etiology (example, viral, fungal, parasitic) during screening or at baseline.
* Participants have signed an informed consent.

Exclusion Criteria:

* Participants with clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial or place the participant at undue medical risk.
* Participants have had a known serious adverse reaction (AR) to immunoglobulin or any anaphylactic reaction to blood or any blood-derived product.
* Participants who have a history of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, diffuse rash, recurrent skin infections, or other disorders where SC therapy would be contraindicated during the study.
* Participants have known isolated IgG subclass deficiency; isolated specific antibody deficiency (SAD) or selective IgG deficiency; or transient hypogammaglobulinemia of infancy.
* Participants have known Selective Immunoglobulin A (IgA) Deficiency (with or without antibodies to IgA).
* Participants have significant proteinuria (≥3+ or known urinary protein loss >1 gram g/24 hours or nephrotic syndrome), has acute renal failure, is on dialysis, and/or has severe renal impairment on Screening laboratory testing (blood urea nitrogen [BUN] or creatinine more than 2.5 times the upper limit of normal [ULN]).
* Participants have screening values of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding more than 2.5 times the ULN for the expected normal range for the testing laboratory.
* Participants have hemoglobin <9 gram per deciliter (g/dL) at screening.
* Participants have a history (either 1 episode within the year prior to the Screening Visit or 2 previous episodes over a lifetime) of or current diagnosis of thromboembolism (example, myocardial infarction, cerebrovascular accident or transient ischemic attack) or deep venous thrombosis.
* Participants are currently receiving anti-coagulation therapy which would make SC administration inadvisable (vitamin K antagonists, nonvitamin K antagonist oral anticoagulants [example, dabigatran etexilate targeting Factor IIa, rivaroxaban, edoxaban, and apixaban targeting Factor Xa], and parenteral anticoagulants [example, fondaparinux]).
* Participants currently have a known hyperviscosity syndrome.
* Participants have an acquired medical condition that is known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000/microliter (μL) [1.0 x10^9/L]), or human immunodeficiency virus infection/acquired immune deficiency syndrome.
* Participants have a known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus or hepatitis C virus infection.
* Participants are receiving any of the following medications: (a) immunosuppressants including chemotherapeutic agents; (b) immunomodulators; (c) long-term systemic corticosteroids defined as daily dose >1 mg of prednisone equivalent/kg/day for >30 days. Note: Intermittent courses of corticosteroids of not more than 10 days would not exclude a participant. Inhaled or topical corticosteroids are allowed.
* Participants (if <18 years of age) have non-controlled arterial hypertension at a level of greater than or equal to the 90th percentile blood pressure (either systolic or diastolic) for their age and height or the adult participant has non-controlled arterial hypertension (systolic blood pressure [SBP] >160 millimeter per mercury (mmHg) and/or diastolic blood pressure [DBP] >100 mmHg).

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Research Solutions of Arizona, PC, Litchfield Park, Arizona
  - Allergy Associates of The Palm Beaches, North Palm Beach, Florida
  - Allergy & Asthma Clinics of Georgia, P.C., Albany, Georgia
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Optimed Research LTD, Columbus, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospect Clinical Research Institute, Tulsa, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - AARA Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with primary immunodeficiency were enrolled at 15 investigative centers in the United States from 24 November 2020 to 25 July 2022.
Period: Overall Study
Arm/Group | IGSC 20%: Treatment-experienced Cohort | IGSC 20%: Treatment-naïve Cohort
Started | 27 | 6
Safety Population (Safety population included all participants who received at least 1 dose of IGSC 20%.) | 27 | 6
Efficacy Evaluable Population (Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.) | 27 | 6
IgG Population (IgG population included all participants who received at least 1 dose of IGSC 20%.) | 27 | 6
Pharmacokinetic (PK) Population (PK population included all the participants who had sufficient PK concentration data to have at least one of the PK parameters: area under the concentration time curve (AUC) (0-7 days), maximum concentration (Cmax), or time to reach Cmax (Tmax).) | 25 | 0
Completed | 24 | 5
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of IGSC 20%.
Groups:
- IGSC 20%: Treatment-experienced Cohort: Participants first received 16 weekly doses of IGSC 20% using a SC infusion pump from Week 0 to Week 15. Participants entering study on IVIG, IGSC 20% was dosed at 1.37 times the equivalent weekly dose and participants entering on SCIG received the same mg/kg equivalent weekly dose as given prior to study entry, without using a DAF. Participants then received 9 biweekly doses of IGSC 20 % (i.e, IGSC 20% every 2 weeks) using an SC infusion pump, with the first IGSC 20% dose administered at Week 16 and the final dose given at Week 32.
- Total: Total of all reporting groups
Arm/Group | IGSC 20%: Treatment-experienced Cohort | IGSC 20%: Treatment-naïve Cohort | Total
Number analyzed (Participants) | 27 | 6 | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 51.7 (12.06) | 56.0 (8.25) | 52.5 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 20
  Male | 11 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 6 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment-experienced Cohort: AUC of IGSC 20% Administered Weekly Assessed as: Steady-State AUC of Total IgG Over a Regular Dosing Interval (τ)
Description: Area under the concentration vs. time curve at steady state over the dosing interval (from time 0 to τ), was calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method was used for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations. The dose interval τ was 7 days for participants on weekly IGSC 20% dosing. The data is reported for participants who received weekly dosing.
Time Frame: Predose and post dose at multiple time points after end of infusion up to Week 15
Population: PK population included all the participants who had sufficient PK concentration data to have at least one of the PK parameters AUC (0-7 days), Cmax, or Tmax. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*milligrams per deciliter (h*mg/dL)
Groups:
- IGSC 20%: Weekly Dosing: Participants received 16 weekly doses of IGSC 20% from Week 0 to Week 15 using a SC infusion pump. Participants entering study IVIG, IGSC 20% was dosed at 1.37 times the equivalent weekly dose and participants entering on SCIG received the same mg/kg equivalent weekly dose as given prior to study entry, without using a DAF.
Arm/Group | IGSC 20%: Weekly Dosing
Number analyzed (Participants) | 23
hours*milligrams per deciliter (h*mg/dL) | 167045.65 (20.2)

2. Primary Outcome: Treatment-experienced Cohort: AUC of IGSC 20% Administered Biweekly Assessed as Steady-State AUC of Total IgG Over a Biweekly Dosing Interval
Description: Area under the concentration vs. time curve at steady state over the dosing interval (from time 0 to τ), was calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method was used for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations. The dose interval τ was 14 days for participants on a biweekly IGSC 20% dosing. AUC (0-14 days) for the biweekly dosing were divided by 2 for comparison with AUC(0-7 days) for the weekly dosing prior to the statistical comparison. The data is reported for participants who received bi-weekly dosing.
Time Frame: Predose and post dose at multiple timepoints after end of infusion up to Week 32
Population: PK population included all the participants who had sufficient PK concentration data to have at least one of the PK parameters AUC (0-7 days), Cmax, or Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mg/dL
Groups:
- IGSC 20%: Bi-Weekly Dosing: Participants received 9 biweekly doses of IGSC 20 % (i.e., IGSC 20% every 2 weeks) using an SC infusion pump, with the first IGSC 20% dose administered at Week 16 and the final dose given at Week 32.
Arm/Group | IGSC 20%: Bi-Weekly Dosing
Number analyzed (Participants) | 23
h*mg/dL
  AUC (0-7 days) | 170926.08 (21.1)
  AUC (0-14 days) | 341852.17 (21.1)
Statistical Analysis 1: Comparison: IGSC 20%: Bi-Weekly Dosing; Geometric least-squares means (GLSMs), GLSM ratio, and 90% CI of GLSM ratio were determined from a mixed-effect model for the log-transformed parameter value with treatment period (weekly or bi-weekly) as a fixed effect and participant as a random effect; Test type: Non-Inferiority — The bi-weekly treatment was considered non-inferior to the weekly treatment if the lower bound of the 90% CI was > 0.8; GLSM Ratio = 1.035, 90% CI 2-sided [1.0030 to 1.0685]

3. Secondary Outcome: Treatment-experienced Cohort: Cmax of Total IgG at Steady State Following IGSC 20% Weekly and Biweekly Administration
Description: The observed maximum total IgG concentration following drug infusion obtained directly from the experimental data without interpolation. The data is reported for participants who received weekly and bi-weekly dosing
Time Frame: Predose and post dose at multiple timepoints after end of infusion up to Week 32
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per deciliter (mg/dL)
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing
Number analyzed (Participants) | 25 | 23
milligrams per deciliter (mg/dL) | 1054.34 (20.6) | 1127.09 (21.4)

4. Secondary Outcome: Treatment-experienced Cohort: Tmax of Total IgG at Steady State Given IGSC 20% Weekly and Biweekly
Description: The data is reported for participants who received weekly and bi-weekly dosing
Time Frame: Predose and post dose at multiple timepoints after end of infusion up to Week 32
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing
Number analyzed (Participants) | 25 | 23
hours | 93.650 [0.00 to 123.03] | 96.233 [71.12 to 264.73]

5. Secondary Outcome: Treatment-experienced Cohort: Steady-State Mean Trough Concentration of Total IgG Following IGSC 20% Weekly and Biweekly Administration
Description: Mean Trough was calculated as the average of the trough concentrations at Weeks 12, 14 Pre-infusion, and 16 for the Weekly Period; and at Weeks 28, 30 Pre-infusion, and 32 for the Biweekly Period. Mean Trough for a given period was not calculated if at least one trough measure was missing. The data is reported for participants who received weekly and bi-weekly dosing.
Time Frame: Predose and post dose at multiple timepoints after end of infusion up to Week 32
Population: IgG population included all participants who received at least 1 dose of IGSC 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing
Number analyzed (Participants) | 27 | 25
mg/dL | 978.29 (18.3) | 960.53 (20.0)
Statistical Analysis 1: Comparison: IGSC 20%: Bi-weekly Dosing; GLSMs, GLSM ratio, and 90% CI of GLSM ratio were determined from a mixed-effect model for the log-transformed parameter value with treatment period (weekly or bi-weekly) as a fixed effect and participants as a random effect; Test type: Non-Inferiority — The biweekly treatment was considered non-inferior to the weekly treatment if the lower bound of the 90% CI was > 0.8; GLSM Ratio = 0.970, 90% CI 2-sided [0.9447 to 0.9957]

6. Secondary Outcome: Treatment-experienced Cohort: Individual Trough Concentration of Total IgG Following IGSC 20% Weekly and Biweekly Administration
Description: IgG Trough 2 = For treatment-experienced participants entering the study on IVIG or Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase (HYQVIA), a second IgG trough level was obtained after screening; this was summarized in the visit designated as IgG Trough 2. Week 0 = Participants entering IVIG or HYQVIA, the first IGSC 20% dose was approximately 1 week post last IVIG/HYQVIA dose and so IgG at Week 0 for these participants represented a pre-dose value. For participants entering on all other forms of SCIG, the Week 0 value is true trough.
Time Frame: Screening, IgG Trough 2, Weeks 0, 2, 4, 8, 12, 14 (pre-infusion), 15, 16, 20, 24, 28, 30 (pre-infusion) and 32
Population: IgG population included all participants who received at least 1 dose of IGSC 20%. Number analyzed is the number of participants with data available for analysis at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | IGSC 20%: Treatment-experienced Cohort
Number analyzed (Participants) | 27
mg/dL
  Screening | 954.7 (24.4)
  IgG Trough 2: number analyzed (Participants) | 9
  IgG Trough 2 | 825.7 (21.5)
  Week 0 | 1071.8 (24.1)
  Week 4: number analyzed (Participants) | 26
  Week 4 | 1069.9 (19.6)
  Week 8: number analyzed (Participants) | 25
  Week 8 | 1052.7 (17.9)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 1012.0 (18.7)
  Week 14: number analyzed (Participants) | 24
  Week 14 | 936.3 (19.2)
  Week 15: number analyzed (Participants) | 24
  Week 15 | 945.0 (19.4)
  Week 16: number analyzed (Participants) | 25
  Week 16 | 1002.1 (18.0)
  Week 20: number analyzed (Participants) | 25
  Week 20 | 952.0 (19.9)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 985.6 (19.8)
  Week 28: number analyzed (Participants) | 23
  Week 28 | 978.8 (22.4)
  Week 30: number analyzed (Participants) | 24
  Week 30 | 933.8 (20.4)
  Week 32 (End of Treatment): number analyzed (Participants) | 24
  Week 32 (End of Treatment) | 966.6 (19.1)

7. Secondary Outcome: Treatment-naïve Cohorts: Individual Trough Concentration of Total IgG
Description: Week 0 = Participants entering IVIG or HYQVIA, the first IGSC 20% dose was approximately 1 week post last IVIG/HYQVIA dose and so IgG at Week 0 for these participants represented a pre-dose value. For participants entering on all other forms of SCIG, the Week 0 value is true trough.
Time Frame: Screening, Weeks 0, 1, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28 and 32
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 6
mg/dL
  Screening | 201.2 (99.9)
  Week 0 | 183.3 (96.7)
  Week 1 | 957.5 (29.1)
  Week 2 | 856.5 (33.1)
  Week 4: number analyzed (Participants) | 5
  Week 4 | 875.3 (25.7)
  Week 6 | 843.5 (22.2)
  Week 8 | 879.1 (24.0)
  Week 10 | 902.4 (20.8)
  Week 12 | 946.2 (18.7)
  Week 16 | 953.9 (16.2)
  Week 20 | 933.7 (21.3)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 938.6 (12.1)
  Week 28: number analyzed (Participants) | 5
  Week 28 | 955.5 (15.1)
  Week 32 (End of Treatment): number analyzed (Participants) | 4
  Week 32 (End of Treatment) | 930.6 (19.5)

8. Secondary Outcome: Treatment-experienced and Treatment-naïve Cohorts: Number of Participants With Serious Bacterial Infection (SBI)
Time Frame: From screening up to final follow up visit at Week 33
Population: Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Measure: Count of Participants; unit: Participants
Arm/Group | IGSC 20%: Treatment-experienced Cohort | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 27 | 6
Participants | 0 | 0

9. Secondary Outcome: Treatment-experienced and Treatment-naïve Cohorts: Rate of Events Per Participant Per Year With Infections of Any Kind as Determined by the Investigator
Description: Rate of events per participant per year was calculated as the total number of events divided by the total duration of exposure in years across all participants. All infections of any kind included serious/nonserious including acute sinusitis, exacerbation of chronic sinusitis, acute otitis media, pneumonia, acute bronchitis, infectious diarrhea etc.) as determined by the investigator. The data is reported for participants in the treatment-naive cohort and the participants who received weekly and bi-weekly dosing.
Time Frame: From screening up to final follow up visit at Week 33
Population: Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Measure: Number (95% Confidence Interval); unit: rate of events per participant per year
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-Weekly Dosing | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 27 | 25 | 6
rate of events per participant per year | 2.299 [1.203 to 4.389] | 1.995 [1.033 to 3.858] | 2.507 [1.198 to 5.247]

10. Secondary Outcome: Treatment-experienced and Treatment-naïve Cohorts: Rate of Events Per Participant Per Year With Validated Infections
Description: Rate of events per participant per year was calculated as the total number of events divided by the total duration of exposure in years across all participants. A validated treatment-emergent infection was documented by positive radiograph, fever (>38°C oral or >39°C rectal), culture, or diagnostic testing for microorganisms e.g., bacterial, viral, fungal, or protozoal pathogens (e.g., rapid streptococcal antigen detection test). Treatment-emergent infection was defined as an infection with onset on or after first infusion start date/time. The data is reported for participants in the treatment-naive cohort and the participants who received weekly and bi-weekly dosing.
Time Frame: From screening up to final follow up visit at Week 33
Population: Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Measure: Number (95% Confidence Interval); unit: rate of events per participant per year
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 27 | 25 | 6
rate of events per participant per year | 0.511 [0.210 to 1.244] | 0.587 [0.213 to 1.615] | 0.279 [0.054 to 1.427]

11. Secondary Outcome: Treatment-experienced and Treatment-naïve Cohorts: Rate of Days Per Participant Per Year That Participants Were on Antibiotics
Description: Rate of days per person per year is calculated as the total number of days divided by the total duration of exposure in years across all participants. Antibiotics included prophylactic and therapeutic. The data is reported for participants in the treatment-naive cohort and the participants who received weekly and bi-weekly dosing.
Time Frame: From screening up to final follow up visit at Week 33
Population: Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Measure: Number (95% Confidence Interval); unit: rate of days per participant per year
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 27 | 25 | 6
rate of days per participant per year
  Prophylactic Antibiotics | 15.326 [5.975 to 39.278] | 15.258 [6.035 to 38.603] | 0.00 [0.000 to NA] — Upper limit of 95% CI was not evaluable due to insufficient number of participants with events.
  Therapeutic Antibiotics | 19.796 [10.493 to 37.316] | 10.681 [5.241 to 21.779] | 23.120 [8.313 to 64.323]

12. Secondary Outcome: Treatment-experienced and Treatment-naïve Cohorts: Rate of Hospitalizations Per Participant Per Year Due to Infection
Description: Rate of hospitalizations per participant per year was calculated as the total number of events divided by the total duration of exposure in years across all participants. Hospitalization was considered only in cases of hospital admission (including emergency room stay) for equal or more than 24 hours. The data is reported for participants in the treatment-naive cohort and the participants who received weekly and bi-weekly dosing.
Time Frame: From screening up to final follow up visit at Week 33
Population: Efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Measure: Number (95% Confidence Interval); unit: rate of events per participant per year
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing | IGSC 20%: Treatment-naïve Cohort
Number analyzed (Participants) | 27 | 25 | 6
rate of events per participant per year | 0.128 [0.048 to 0.340] | 0.117 [0.043 to 0.323] | 0.000 [0.000 to NA] — Upper limit of 95% CI was not evaluable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From screening up to final follow up visit at Week 33
Description: Safety population included all participants who received at least 1 dose of IGSC 20%. The data for all-cause mortality, serious adverse events, and non-serious adverse events is reported for participants in the treatment-naive cohort and the participants who received weekly and bi-weekly dosing.
Arm/Group | IGSC 20%: Weekly Dosing | IGSC 20%: Bi-weekly Dosing | IGSC 20%: Treatment-naïve Cohort
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/25 | 1/6
Other Adverse Events (participants affected / at risk) | 4/27 | 1/25 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC 20%: Weekly Dosing (N=27) | IGSC 20%: Bi-weekly Dosing (N=25) | IGSC 20%: Treatment-naïve Cohort (N=6)
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC 20%: Weekly Dosing (N=27) | IGSC 20%: Bi-weekly Dosing (N=25) | IGSC 20%: Treatment-naïve Cohort (N=6)
Headache (Nervous system disorders) | 3 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Infusion site reaction (General disorders) | 0 | 0 | 1
Infusion site scab (General disorders) | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study after 12 months of study completion date or after Grifols confirms there will be no joint, multi-center publication, then institution and/or investigator shall have the right, at their discretion, to publish, either in writing or orally, the results of the study performed under the protocol under certain conditions. At Sponsors' request, Site will remove any Confidential Information (other than Study results).

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04566692/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04566692/SAP_001.pdf